CLINICAL TRIAL: NCT02621736
Title: Copeptin for Prediction of Treatment Response in Children With Monosymptomatic Nocturnal Enuresis (MEN).
Acronym: COMEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: EK 2015-340
Record Dates: First submitted 2015-11-25; First posted 2015-12-03 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Nocturnal Enuresis
Keywords: children; desmopressin; copeptin
MeSH Terms: conditions — Nocturnal Enuresis; Diabetes Insipidus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood sampling — At 4 visits capillary blood sampling for copeptin measurement will be performed with each child.

SUMMARY:
Monosymptomatic nocturnal enuresis (MEN) is a common problem in children, affecting 7-10% of all 7 year olds. MEN is often leading to psychosocial problems because of its burden and stigmatism.

The only available medical treatment option is the vasopressin analogum Desmopressin®. However, according to the literature, only one third of patients shows a good treatment response, defined as more than 90% of reduced bed wetting. Furthermore, treatment with Desmopressin® may lead to psychosocial problems, high costs and potentially dangerous side effects like water intoxication and hypertension.

Copeptin, mirroring arginine vasopressin (AVP), has been shown to be significantly lower in patients with MEN compared to controls and lower in patients with severe bed wetting compared to patients with only slight bed wetting.

ELIGIBILITY:
Inclusion Criteria:

* Children at the age between 5 and 16 years
* Diagnosis of monosymptomatic nocturnal enuresis
* Completion of uroflowmetry and bladder sonography if possible
* Completion of home recording charts of bed wetting episodes if possible
* Willingness to use Desmopressin® treatment

Exclusion Criteria:

* Children with daytime enuresis
* Children with lower urinary tract symptoms and infection
* Children with structural abnormalities of the urinary tract
* Children with chronic illness, esp. renal failure, hypertension, congenital heart disease, diabetes mellitus and diabetes insipidus.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children at the Age of 5-16 years with monosymptomatic enuresis nocturna
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change of copeptin at baseline and after 28 days during routine desmopressin therapy | morning and evening copeptin levels at baseline day 0 before routine desmopressin therapy and day 28 during routine desmopressin therapy

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Professor, Principal Investigator — University Hospital Basel, Department of Endocrinology, Diabetes and Metabolism
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No